CLINICAL TRIAL: NCT03997058
Title: The First Affiliated Hospital of Guangzhou University of Chinese Medicine
Brief Title: Observation on the Effect of Auricular Acupoint Pressing on Insomnia and Adverse Events in MHD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Haitao Tu, Principal Investigator, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191114
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Renal Dialysis; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Negative control group, auricular acupoint pressing group, estazolam group， combined treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention)
- Auricular acupoint pressing group (Experimental)
  Interventions: Other: Auricular point pressure therapy
- Oral estazolam group (Active Comparator)
  Interventions: Drug: Oral estazolam medication
- Combined treatment group (Active Comparator)
  Interventions: Other: Auricular point pressure therapy; Drug: Oral estazolam medication

INTERVENTIONS:
Other: Auricular point pressure therapy — Use a hard and smooth pill to adhere to the center of the 0.7×0.7cm tape. Hold the puncture clip on the part of the ear which is selected, and give appropriate pressure (揉) to make the patient have heat, hemp, Swelling and painful feeling; patients with sputum press 3-5 times a day, each time 1-2 minutes per hole, and must be pressed once every 15-30 minutes before going to bed every night. Press the point pressure method (press the ear point with a fingertip and press it loosely, each interval is 0.5 seconds. It is better for the patient to feel the swelling and slightly heavy tingling, and the force should not be too heavy. Generally, each time the hole can be pressed 27 times. Each time one side of the ear is selected, the two ear points are used alternately, staying in the summer for 1-3 days, and staying in the winter for 3-7 days.It is not appropriate to have local inflammation of the auricle, frostbite or surface skin ulceration.
  Arms: Auricular acupoint pressing group; Combined treatment group
Drug: Oral estazolam medication — The first dose was started from 0.5mg, qn, and taken at 30min-1h before going to bed. If the dose is not effective, gradually increase the amount to 2mg, qn. If the patient has drug-induced liver damage and respiratory depression, it is necessary to stop the drug immediately. Hemorrhoids avoid drinking alcohol during medication.
  Arms: Combined treatment group; Oral estazolam group

SUMMARY:
Maintenance hemodialysis (MHD) is one of the most important treatments for patients with end-stage renal failure. Studies have found that insomnia is widespread in MHD patients, affecting their quality of life. Auricular acupoint pressing is an effective traditional Chinese medicine treatment for insomnia. This study compared the effects of auricular acupoint pressing and oral estazolam on insomnia in patients with MHD, and evaluated the possibility of auricular acupoint pressing to reduce the incidence of adverse events by improving insomnia in patients with MHD, and to explore the insomnia of MHD patients treated with TCM characteristics. The role and efficacy provide a basis for the treatment of sleep disorders by Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

1.Age 18-90 years old，received maintenance hemodialysis treatment for more than 1 year, no history of surgical trauma, infection, trauma in the past 3 months; 2.the current condition is stable, the heart function is grade I, no limb paralysis, speech disadvantages and other sequelae； 3.Informed consent volunteer to participate in this experiment.

Exclusion Criteria:

1. At present, dialysis is inadequate, water and sodium retention is severe;
2. combined with severe cardiovascular disease, sequelae of cerebral infarction or history of cerebral hemorrhage, history of COPD, history of myasthenia gravis, history of angle-closure glaucoma, blood system disease, mental system disease or other systemic The disease can not be matched with the experimenter;
3. poor compliance or poor medical attitude;
4. severe hearing or vision loss, or a very low level of education, can not match the experiment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index（PSQI）score | June 1, 2019 to June 1, 2021
Mortality rate | June 1, 2019 to June 1, 2021

SECONDARY OUTCOMES:
Incidence of cardiovascular events | June 1, 2019 to June 1, 2021
Cerebrovascular accident rate | June 1, 2019 to June 1, 2021
Gastrointestinal bleeding rate | June 1, 2019 to June 1, 2021

OTHER OUTCOMES:
Hypersensitive C-reactive protein concentration | June 1, 2019 to June 1, 2021

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzho University of Chinese Medicine, Guangzhou, Guangdong, China